CLINICAL TRIAL: NCT00522665
Title: Phase I / Randomized Phase II Study of Second Line Therapy With Irinotecan and Cetuximab With or Without RAD001, an Oral mTOR Inhibitor for Patients With Metastatic Colorectal Cancer: Hoosier Oncology Group GI05-102
Brief Title: Phase I/Randomized Phase II Study of Second Line Therapy With Irinotecan + Cetuximab +/- RAD001 for Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GI05-102
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Cetuximab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Irinotecan + Cetuximab +/- RAD001 (Active Comparator)
  Interventions: Drug: Irinotecan; Biological: Cetuximab; Biological: RAD001
- Arm B: Ironotecan + Cetuximab (Active Comparator)
  Interventions: Drug: Irinotecan; Biological: Cetuximab

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 125 mg/m2 IV days 1 and 8
Biological: Cetuximab — Cetuximab 250mg/m2 IV days 1, 8 and 15
Biological: RAD001 — Patients on Arm A will crossover and receive RAD001 at disease progression
  Arms: Arm A: Irinotecan + Cetuximab +/- RAD001

SUMMARY:
The addition of RAD001, an mTOR inhibitor, to irinotecan and anti-EGFR antibody cetuximab may increase efficacy for patients with metastatic colorectal cancer who progressed on prior chemotherapy. This approach is biologically directed to overall target the cancer cell at multiple levels, and potentially preventing chemotherapy and EGFR-therapy resistance.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

PHASE I:

* UGT1A1 *28 7/7 genotype IS NOT present
* Cetuximab 250 mg/m2 IV days 1, 8, and 15
* Irinotecan 125 mg/m2 IV days 1 and 8
* RAD001 PO QD (dose determined at the time of registration; subjects will remain at this dose level until treatment discontinuation)

PHASE II:

* Randomization based on UGT1A1 *28 7/7 Genotype or Prior Irinotecan Exposure

ARM A:

* Cetuximab 250 mg/m2 IV days 1, 8, and 15
* Irinotecan 125 mg/m2 IV days 1 and 8

AT TIME OF PROGRESSIVE DISEASE, ARM A TREATMENT WILL CROSSOVER:

* Cetuximab 250 mg/m2 IV days 1, 8, and 15
* Irinotecan 125 mg/m2 IV days 1 and 8
* RAD001 PO QD (maximum tolerated dose)

ARM B:

* Cetuximab 250 mg/m2 IV days 1, 8, and 15
* Irinotecan 125 mg/m2 IV days 1 and 8
* RAD001 PO QD (maximum tolerated dose)

AT TIME OF PROGRESSIVE DISEASE, ARM B TREATMENT WILL BE DISCONTINUED

ECOG performance status 0-2

Life Expectancy: Not specified

Hematopoietic:

* Absolute neutrophil count (ANC) ≥ 1,500 mm3
* Platelets ≥ 100,000 mm3
* Hemoglobin (Hgb) ≥ 9 g/dL
* White blood cell count (WBC) ≥ 2,000 mm3
* INR < 1.5 x upper limit of normal (ULN) if not on anticoagulation (if on anticoagulation must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin)
* PTT < 1.5 x ULN

Hepatic:

* Bilirubin ≤ 1.5 x ULN
* Aspartate aminotransferase (AST, SGOT) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT, SGPT) ≤ 2.5 x ULN
* Albumin ≥ 3.0 g/dL

Renal:

* Calculated creatinine clearance of ≥ 60 cc/min using the Cockcroft-Gault formula

Cardiovascular:

* No uncontrolled cardiac arrhythmia requiring medication, transient ischemic attack (TIA), or cerebrovascular accident (CVA) within 6 months prior to being registered for protocol therapy
* No uncontrolled congestive heart failure, myocardial infarction, or unstable angina within 6 months prior to being registered for protocol therapy

Pulmonary:

* No severely impaired lung function as demonstrated by pulse O2 saturation ≤ 90% at rest on room air, or pulmonary function test FEV1 ≤ 2L
* No history of prior chronic lung infection such as tuberculosis, atypical tuberculosis, or histoplasmosis as evidenced by a chest CT or x-ray within 21 days prior to being registered for protocol therapy

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of colon or rectal adenocarcinoma
* Measurable site of disease according to RECIST that has not been previously irradiated
* Must have metastatic colorectal cancer which progressed after first line chemotherapy +/- bevacizumab
* Blood sample collected within 21 days prior to being registered for protocol therapy for UTG1A1 genotype analysis. (Patients with the UGT1A1 *28 7/7 genotype (homozygosity for the TA7 allele) will be excluded from the Phase I stage of the study. During the Phase II stage of the study, subjects will be allowed to participate but must begin treatment at dose level -1 of irinotecan.)
* A history of other malignancies (non-colorectal) is allowed, provided it has been curatively treated and demonstrates no evidence for recurrence of that cancer
* Prior radiation therapy allowed to < 25% of the bone marrow
* Age ≥ 18 years at the time of consent
* Written informed consent and HIPAA authorization for release of personal health information
* Females of childbearing potential and males must be willing to use an effective method of contraception
* Females of childbearing potential must have a negative pregnancy test within 7 days of being registered for protocol therapy

Exclusion Criteria:

* No more than one prior chemotherapy regimen for metastatic colorectal cancer, at least 28 days prior to being registered for protocol therapy
* No prior treatment with cetuximab
* No prior treatment with an mTOR inhibitor
* No known hypersensitivity to cetuximab, RAD001 (everolimus), other rapamycins (sirolimus, temsirolimus) or to its excipients
* No treatment with any investigational agent within 28 days prior to being registered for protocol therapy
* No symptomatic brain metastasis
* No uncontrolled diabetes as defined by a fasting serum glucose >1.5 x ULN
* No chronic treatment with systemic steroids or another immuno-suppressive agent
* No serious non-healing wound, ulcer, bone fracture, major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to being registered for protocol therapy
* No liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* No active bleeding or a pathological condition that is associated with a high risk of bleeding
* No uncontrolled systemic disease including active infections or uncontrolled hypertension
* No known history of HIV seropositivity
* No impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* No nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with protocol therapy
* No planned immunization with attenuated live viruses during the study period
* Females must not be breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2011-05 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To determine the MTD of RAD001 in combination with irinotecan and cetuximab as second line therapy in patients with metastatic colorectal cancer | Phase I
To evaluate the objective response (CR or PR) rates of patients treated with irinotecan and cetuximab with or without RAD001 in patients with metastatic colorectal cancer | Phase II

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic (PK) profile for RAD001 after one cycle of therapy, on cycle 2 day 1 | Phase I
To evaluate the time to progression, duration of objective response (CR or PR) and overall survival of patients treated with irinotecan and cetuximab with or without RAD001 | Phase II

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Chiorean, M.D., Study Chair — Hoosier Oncology Group, Inc.
Locations (14):
- United States (14):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - IN Onc/Hem Associates, Indianapolis, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Hospital & Health Centers, Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - Center for Cancer Care, Inc., P.C., New Albany, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Siteman Cancer Center, St Louis, Missouri

REFERENCES:
- [Result] Chiorean EG, Picus J, Breen T, Ansari RH, Harb WA, Burns M, Spittler AJ, Loehrer PJ. Phase I/II study of everolimus (E) with irinotecan (Iri) and cetuximab (C) in 2nd line metastatic colorectal cancer (mCRC): Hoosier Cancer Research Network GI05-102. J Clin Oncol 33:5s, 2015 (suppl; abstr 3618)
- See also: Hoosier Cancer Research Network Homepage — http://www.hoosiercancer.org